CLINICAL TRIAL: NCT05995964
Title: A PHASE 2, RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED STUDY TO INVESTIGATE THE EFFICACY AND SAFETY OF PF-07275315 AND PF-07264660 IN ADULT PARTICIPANTS WITH MODERATE-SEVERE ATOPIC DERMATITIS
Brief Title: A Study To Learn About Two Study Medicines (PF-07275315 And PF-07264660) In People Who Have Moderate To Severe Atopic Dermatitis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C4531002; 2023-505218-68-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2023-07-26; First posted 2023-08-16 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Atopic Dermatitis
Keywords: Eczema
MeSH Terms: conditions — Dermatitis, Atopic; Eczema

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (14):
- Stage 1_PF-07275315 (Experimental): Stage 1 PF-07275315 Injections over 12 weeks
  Interventions: Drug: PF-07275315
- Stage 1_PF-07264660 (Experimental): Stage 1 PF-07264660 Injections over 12 weeks
  Interventions: Drug: PF-07264660
- Stage 1_Placebo (Experimental): Stage 1 Placebo Injections over 12 weeks
  Interventions: Other: Placebo
- Stage 2_PF-07275315 _Dose A (Experimental): Stage 2 PF-07275315 Injections over 12 weeks.
  Interventions: Drug: PF-07275315
- Stage 2_PF-07275315 _Dose B (Experimental): Stage 2 PF-07275315 Injections over 12 weeks.
  Interventions: Drug: PF-07275315
- Stage 2_PF-07275315 _Dose C (Experimental): Stage 2 PF-07275315 Injections over 12 weeks.
  Interventions: Drug: PF-07275315
- Stage 2_PF-07275315 _Dose D (Experimental): Stage 2 PF-07275315 or PF-07264660 Injections over 12 weeks.
  Interventions: Drug: PF-07275315; Drug: PF-07264660
- Stage 2_Placebo (Experimental): Stage 2 Placebo Injections over 12 weeks.
  Interventions: Other: Placebo
- Stage 3_Placebo+PF-07275315_Dose A (Experimental): Stage 3 Placebo Injections for 16 weeks followed by PF-07275315 Injections for 16 weeks.
  Interventions: Drug: PF-07275315; Other: Placebo
- Stage 3_PF-07275315_Dose B (Experimental): Stage 3 PF-07275315 Injections for 32 weeks.
  Interventions: Drug: PF-07275315
- Stage 4_PF-07264660_Dose A (Experimental): Stage 4 PF-07264660 Injections for 12 weeks
  Interventions: Drug: PF-07264660
- Stage 4_PF-07264660_Dose B (Experimental): Stage 4 PF-07264660 Injections for 12 weeks
  Interventions: Drug: PF-07264660
- Stage 4_PF-07264660_Dose C (Experimental): Stage 4 PF-07264660 Injections for 12 weeks
  Interventions: Drug: PF-07264660
- Stage 4_Placebo (Experimental): Stage 2 Placebo Injections for 12 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: PF-07275315 — subcutaneous injection
  Arms: Stage 1_PF-07275315; Stage 2_PF-07275315 _Dose A; Stage 2_PF-07275315 _Dose B; Stage 2_PF-07275315 _Dose C; Stage 2_PF-07275315 _Dose D; Stage 3_PF-07275315_Dose B; Stage 3_Placebo+PF-07275315_Dose A
Drug: PF-07264660 — subcutaneous injection
  Arms: Stage 1_PF-07264660; Stage 2_PF-07275315 _Dose D; Stage 4_PF-07264660_Dose A; Stage 4_PF-07264660_Dose B; Stage 4_PF-07264660_Dose C
Other: Placebo — subcutaneous injection
  Arms: Stage 1_Placebo; Stage 2_Placebo; Stage 3_Placebo+PF-07275315_Dose A; Stage 4_Placebo

SUMMARY:
The purpose of this study is to learn about the safety and effects of 2 study medicines (PF-07275315 and PF-07264660) for the treatment of atopic dermatitis (AD). AD is a long- lasting itchy red rash, caused by a skin reaction.

This study is seeking participants who:

* are 18 years of age or more.
* Were confirmed to have AD at least 6 months ago.
* Are not having an effective treatment result from medicines that are applied on skin for AD.
* Are considered by their doctors to have moderate to severe AD.

In Stage 1 of the study, participants will receive either PF-07275315 or PF-07264660 or placebo. Stage 1 is complete. In Stage 2 of the study participants will receive either PF-07275315 or placebo. In Stage 3 of the study participants who have received anti-inflammatory proteins, will receive either PF-07275315 or placebo. In Stage 4 of the study participants will receive either PF-07264660 or placebo. A placebo does not have any medicine in it but looks just like the medicines being studied.

PF-07275315 or PF-07264660 or placebo will be given as multiple shots in the clinic over the course of each Stage.

The experiences of people receiving PF-07275315 or PF-07264660 will be compared to people who do not. This will help determine if PF-07275315 and PF-07264660 are safe and effective.

Participants in Stages 1, 2 and 4 will be involved in this study for up to 40 weeks (10 months). Participants in Stage 3 will be involved in this study for up to 52 weeks (13 months).

ELIGIBILITY:
Inclusion Criteria:

Must meet the following AD criteria:

1. Participants aged 18 years or older
2. Clinical diagnosis of chronic atopic dermatitis:

   1. for at least 6 months prior to Day 1 with diagnosis confirmed by photograph;
   2. Either an inadequate response to treatment with standard of care treatments (excluding systemic immunosuppressant treatments) for at least 4 consecutive weeks within 6 to 12 months of the first dose of the study intervention; OR documented reason why topical treatments are considered medically inappropriate;
   3. Moderate to severe AD defined as having an affected BSA ≥10%, vIGA ≥3, and EASI ≥16 at both the screening and baseline visits).
   4. Bio-experienced cohort-partial or non-responder to anti-inflammatory proteins (also known as biologics), intolerance or AEs to anti-inflammatory proteins or loss of access to anti-inflammatory proteins with ≥12 weeks of treatment within 5 years.

   Other Inclusion Criteria:
3. BMI of 17.5 to 40 kg/m2; and a total body weight >45 kg (100 lbs).
4. Willing and able to comply with all scheduled visits, treatment plan, laboratory tests and other study procedures.

Exclusion Criteria:

- Medical Conditions:

1. Significant allergic or autoimmune diseases, other than AD and well controlled mild to moderate including but not limited to: SLE or other complement disorders; Type 1 diabetes; IBD; Multiple Sclerosis.
2. History of significant allergic reactions, including anaphylaxis and reactions to protein therapeutics, including hypersensitivity to PF-07275315 or PF-07264660 or to the excipients of the formulated drug products. Participants with significant reactions to single, identified, avoidable allergens (eg, peanut allergy) may be eligible if avoidance of these allergens during the study is feasible.
3. Any of the following acute or chronic infections or infection history:

   1. Active infection (including helminth or parasitic) requiring treatment within 2 weeks prior to screening;
   2. Infection requiring hospitalization or systemic (parenteral) antimicrobial therapy within 60 days prior to Day 1;
   3. Active chronic or acute skin infection requiring treatment with systemic [(not IV)] antibiotics, antivirals, antiparasitics, antiprotozoals, or antifungals within 2 weeks prior to Day 1, or superficial skin infections (requiring no more than topical anti-infective treatments) within 1 week prior to Day 1.
   4. Any infection judged to be an opportunistic infection or clinically significant by the investigator, within 6 months prior to Day 1;
4. History of or current evidence of inflammatory skin conditions (eg, psoriasis, seborrheic dermatitis, lupus) at the time of Day 1 that could interfere with evaluation of AD or response to treatment.
5. Any medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.

   - Prior/Concomitant Therapy:
6. Current use of any prohibited concomitant medication(s).
7. Phototherapy narrowband UVB (NB UVB) or broadband phototherapy or regular use (more than 2 visits per week) of a tanning booth/parlor within 4 weeks prior to Day 1.

   - Prior/Concurrent Clinical Study Experience:
8. Previous administration with an investigational product (drug or vaccine) within 30 days (or as determined by the local requirement) or 5 half lives preceding the first dose of study intervention used in this study (whichever is longer).
9. HIV infection, or infection with hepatitis B or hepatitis C viruses according to protocol-specific testing algorithm.
10. Evidence of active or latent TB, or inadequately treated infection with Mycobacterium TB. A participant who is currently being treated for active or latent TB infection must be excluded from this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2023-08-22 (Actual); Primary Completion 2026-09-21 (Estimated); Study Completion 2026-12-14 (Estimated)

PRIMARY OUTCOMES:
The number of participants achieving ≥75% improvement in EAS175 from baseline at week16. | Week 16
  EASI75 (≥75% improvement from baseline) at Week 16

SECONDARY OUTCOMES:
The number and % of participants achieving vIGA score of clear (0) or almost clear (1) (on a 5-point scale) and a reduction from baseline of ≥2 points at all scheduled time points | Screening through study completion, an average of 36 weeks.
  vIGA score of clear (0) or almost clear (1) (on a 5-point scale) and a reduction from baseline of ≥2 points at all scheduled time points
The number and % of participants achieving EASI75 (≥75% improvement from baseline) at scheduled time points except Week 16 | All scheduled timepoints other than Week 16, screening through study completion, an average of 36 weeks.
  EASI75 (≥75% improvement from baseline) at scheduled time points except Week 16
The number and % of participants achieving a Percent change from baseline in EASI total score at scheduled time points | Screening through study completion, an average of 36 weeks.
  Percent change from baseline in EASI total score at scheduled time points
The number and % of participants with treatment emergent AEs | Screening - Week 36
  Incidence of treatment emergent AEs
The number and % of participants with clinically significant changes in vital signs | Screening - Week 36
  Incidence of clinically significant changes in vital signs
The number and % of participants with clinically significant changes in ECG | Screening - Week 36
  Incidence of clinically significant changes in ECG
The number and % of participants with clinically significant changes in laboratory tests | Screening - Week 36
  Incidence of clinically significant changes in laboratory tests

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (95):
- United States (52):
  - Allervie Clinical Research, Birmingham, Alabama
  - Onyx Clinical Research - Peoria, Peoria, Arizona
  - Medical Dermatology Specialists, Phoenix, Arizona
  - Onyx Clinical Research, Phoenix, Arizona
  - Banner - University Medicine Dermatology Clinic, Tucson, Arizona
  - Marvel Clinical Research, Huntington Beach, California
  - California Allergy and Asthma Medical Group, Los Angeles, California
  - University Dermatology Trials, INC., Newport Beach, California
  - Northridge Clinical Trials, Northridge, California
  - Profound Research LLC, Oceanside, California
  - Dermatology Cosmetic Laser Medical Associates of La Jolla, Inc., San Diego, California
  - Sunwise Clinical Research, Walnut Creek, California
  - AboutSkin Research, LLC, Greenwood Village, Colorado
  - Renaissance Research and Medical Group, Cape Coral, Florida
  - Florida International Medical Research, Coral Gables, Florida
  - Revival Research, Doral, Florida
  - St. Jude Clinical Research, Doral, Florida
  - SouthCoast Research Center, Miami, Florida
  - Floridian Research Institute Llc, Miami, Florida
  - Global Health Research Center, Inc., Miami Lakes, Florida
  - Ziaderm Research LLC, North Miami Beach, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - GCP Research, Global Clinical professionals, St. Petersburg, Florida
  - ForCare Clinical Research, Tampa, Florida
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - Southern Indiana Clinical Trials, New Albany, Indiana
  - Maryland Laser Skin and Vein, Hunt Valley, Maryland
  - Michigan Center for Research Company, Clarkston, Michigan
  - MI Skin Innovations, Northville, Michigan
  - Revival Research Institute LLC, Troy, Michigan
  - Revival Research Institute, LLC, Troy, Michigan
  - Skin Specialists, PC dba Schlessinger MD, Omaha, Nebraska
  - Empire Dermatology, East Syracuse, New York
  - Private Practice - Dr. Bobby Buka, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Sadick Research Group, New York, New York
  - Apex Clinical Research Center, Mayfield Heights, Ohio
  - Epic Medical Research - Oklahoma, Chickasha, Oklahoma
  - Unity Clinical Research, Oklahoma City, Oklahoma
  - Vital Prospects Clinical Research Institute, PC, Tulsa, Oklahoma
  - Velocity Clinical Research, Medford, Medford, Oregon
  - Paddington Testing Co, Inc, Philadelphia, Pennsylvania
  - Clinical Partners, LLC, Johnston, Rhode Island
  - National Allergy and Asthma, North Charleston, South Carolina
  - Spartanburg Medical Research, Spartanburg, South Carolina
  - Clinical Neuroscience Solutions Inc., Memphis, Tennessee
  - Dermatology Treatment and Research Center, Dallas, Texas
  - North Texas Center for Clinical Research, Frisco, Texas
  - Alpesh D. Desai, DO PLLC, Houston, Texas
  - DCT-Stone Oak, LLC dba Discovery Clinical Trials, San Antonio, Texas
  - Complete Dermatology, Sugar Land, Texas
  - Virginia Dermatology and Skin Cancer Center, Norfolk, Virginia
- Australia (4):
  - Australian Clinical Research Network, Sydney, New South Wales
  - Box Hill Hospital, Box Hill, Victoria
  - Dr Rodney Sinclair Pty Ltd, East Melbourne, Victoria
  - Fremantle Dermatology, Fremantle, Western Australia
- Canada (8):
  - Wiseman Dermatology Research Inc., Winnipeg, Manitoba
  - Medicor Research Inc, Greater Sudbury, Ontario
  - Sudbury Skin Clinique, Greater Sudbury, Ontario
  - Lima's Excellence in Allergy and Dermatology Research, Hamilton, Ontario
  - DermEdge Research, Mississauga, Ontario
  - Toronto Research Centre, Toronto, Ontario
  - INTERMED Groupe Sante, Chicoutimi, Quebec
  - Centre de Recherche Saint-Louis inc., Québec
- China (16):
  - Beijing Friendship Hospital Affiliate of Capital University, Beijing, Beijing Municipality
  - The First Affiliated Hospital Of Fujian Medical University, Fuzhou, Fujian
  - Guangdong Province Dermatology Hospital, Guangzhou, Guangdong
  - The First Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The Second Xiangya Hospital of Central South University, Changsha, Hu'nan
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Dermatology Hospital of Jiangxi Province, Nanchang, Jiangxi
  - The first hospital of jilin university, Changchun, Jilin
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Huashan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Hangzhou Third Hospital, Hangzhou, Zhejiang
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Chengdu second people's hospital, Chengdu
  - Shanghai First People's Hospital, Shanghai
- Germany (3):
  - Fachklinik Bad Bentheim, Bad Bentheim, Lower Saxony
  - BAG Drs. Med. Quist PartG, Mainz, Rhineland-Palatinate
  - Magdeburger Company for Medical Studies and Services, Magdeburg, Saxony-Anhalt
- Japan (6):
  - Nomura Dermatology Clinic, Yokohama, Kanagawa
  - Medical Corporation Heishinkai OPHAC Hospital, Osaka, Osaka
  - Osaka Metropolitan University Hospital, Osaka, Osaka
  - Nihonbashi Sakura Clinic, Chuo-ku, Tokyo
  - Fukuwa Clinic, Chuo-ku, Tokyo
  - Naoko Dermatology Clinic, Setagaya-ku, Tokyo
- Poland (6):
  - Niepubliczny Zakład Opieki Zdrowotnej Zespół Poradni Specjalistycznych "Termedica", Poznan, Greater Poland Voivodeship
  - Pratia MCM Krakow, Krakow, Lesser Poland Voivodeship
  - Synexus Polska Sp. z o.o. Oddzial we Wroclawiu, Wroclaw, Lower Silesian Voivodeship
  - Centrum Medyczne Angelius Provita, Katowice, Silesian Voivodeship
  - Synexus Polska Sp. z o.o. Oddzial w Katowicach, Katowice
  - Dermedic Jacek Zdybski, Ostrowiec Świętokrzyski, Świętokrzyskie Voivodeship

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4531002